CLINICAL TRIAL: NCT03858920
Title: The Liver in the World Trade Center Health Program General Responder Cohort and Controls
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Andrea Branch, Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 16-2612; U01OH011489-01 (NIH); IF 1991038 (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2018-02-27; First posted 2019-03-01 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Steatosis of Liver; NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- General Responder Cohort (GRC) WTC Responders: General Responder Cohort (GRC) and who have chosen to undergo annual medical monitoring and treatment of their WTC-related conditions at Mount Sinai's Irving J. Selikoff Center for Occupational and Environmental Medicine (SCOEM), which is directed by Dr. M. Crane
  Interventions: Device: Fibroscan of Liver; Procedure: Low-dose non-contrast CT
- General Responder Cohort (GRC) Non WTC Responders: Members of the World Trade Center General Non Responder Cohort.
  Interventions: Device: Fibroscan of Liver; Procedure: Low-dose non-contrast CT

INTERVENTIONS:
Device: Fibroscan of Liver — A non-invasive diagnostic device used to measure liver scarring
  Other Names: FibroScan Test
Procedure: Low-dose non-contrast CT — CT scan as part of routine research care

SUMMARY:
This project investigates whether exposure to the World Trade Center Attack is a risk factor for liver injury.

DETAILED DESCRIPTION:
This is a prospective cross-sectional study of liver disease in individuals who meet the United States Preventive Services Task Forces guidelines for lung cancer screening because they are between 55 and 80 years of age and have a 30 year pack-history of smoking and are either current smokers or who quit during the past 15 years. Liver disease will be compared between individuals who are members of the World Trade Center General Responder Cohort and individuals who are not members of this cohort. The basic objective is to determine whether exposure to the WTC attack increased liver disease.

Data will be obtained from the World Trade Center Data Center, from Mount Sinai Medical records, EPIC, the data warehouse, and from data collected by the Lung Cancer Screening Program of Dr. Henschke. Results of genetic tests that relate to liver disease will be collected from the medical record.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female between 55 and 80 years of age
* 30 year pack-history of smoking and are either current smokers or who quit during the past 15 years.
* Individuals who are members of the World Trade Center General Responder Cohort or Subjects who meet the United States Preventive Services Task Forces guidelines for lung cancer screening

Exclusion Criteria:

* None

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Members of the World Trade Center General Responder Cohort and individuals who are not members of this cohort.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
FibroScan- Controlled Attenuation Parameter (CAP) scores | Day 1
  assesses liver fat using a patented technique called Vibration-Controlled Transient Elastography range from 0 -400 CAP with the higher number indicating great quantity of fat in the Liver CAP 240-270 S1 Mild Steatosis CAP 270-300 S2 Moderate Steatosis CAP >300 S3 Severe Steatosis
Attenuation Hounsfeld units signal intensity in low -dose non-contrast CT scan | Day 1
  The attenuation of Hounsfeld units (HU) signal intensity in low-dose non-contrast CT to estimate liver fibrosis
Fibroscan | Day 1
  assesses liver stiffness using a patented technique called Vibration-Controlled Transient Elastography. Results are measured using kiloPascal's (or kPa) and range from 2 to 75kPa, with a higher number indicating more liver scarring.
  F0 Zero 5.3 kPa means no scarring F1 5.3-7.0 kPa is mild fibrosis F2 is 7.1-8.0 kPa moderate fibrosis F3 8.1-12.4 kPa is severe fibrosis F4 greater than 12.5 kPa is cirrhosis or advanced fibrosis,

SECONDARY OUTCOMES:
Relationship between WTC exposure and liver fat | Day 1
  The Controlled Attenuation Parameter (CAP) scores using a Multiple linear regression modeling to determine whether WTC exposure is significantly associated with liver fat content after adjusting for potential confounding factors ,smoking history, diabetes and BMI.
Composite score for Fibrosis and Steatosis | Day 1
  Composite score from Fibroscan to compare for exposure to WTC site Clinically significant fibrosis will be defined as Fibroscan >8.0kPa and Steatosis will be defined as a Fibroscan CAP >300dB/m indicating advance steatosis <7.9 kPa score Zero , >8.0 kPa score 1, <299 CAP will score Zero, >300 CAP will score 1 Range of total score Zero -2 equals best to worst scoring

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Branch, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided